CLINICAL TRIAL: NCT03821844
Title: Music & MEmory: A Pragmatic TRial for Nursing Home Residents With ALzheimer's Disease_part1
Acronym: METRIcAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Westat (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Vincent Mor, Florence Pirce Grant University Professor, Professor of Health Services, Policy and Practice, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R33AG057451_part1; R33AG057451 (NIH)
Record Dates: First submitted 2018-10-18; First posted 2019-01-30 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The investigator's primary outcome (staff report of resident agitated and aggressive behaviors) will be evaluated using a parallel design. Some secondary outcomes will be tested with a stepped wedge design.
Who Masked: Investigator
Masking Description: The principal investigator is blinded to random assignment of nursing homes to treatment or control conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music and Memory (Experimental): Music and Memory is a personalized music program in which nursing home staff provide people with dementia with music playlists tailored to their personal history of music preferences.
  Interventions: Behavioral: Music and Memory
- Usual Care (No Intervention): Usual care for managing agitated and/or aggressive behaviors in the nursing home setting.

INTERVENTIONS:
Behavioral: Music and Memory — Music and Memory is a personalized music program in which caregivers (nursing home staff, family, or others) provide people with dementia with music playlists tailored to their personal history of music preferences.
  Arms: Music and Memory

SUMMARY:
The purpose of this trial is to test the effects of a personalized music intervention (Music and Memory, Inc.) on agitated and aggressive behaviors for nursing home residents with dementia.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a parallel, pragmatic, cluster randomized control trial of personalized music (Music and Memory) for nursing home residents with moderate to severe dementia living in 54 nursing homes (27 treatment, 27 control) from 4 nursing home corporations. Music and Memory is a personalized music program that uses portable music players to deliver individualized music to people with dementia at times when agitated behaviors are likely.

**This funding mechanism sponsored two parallel trials with different implementation strategies. In this trial, nursing home staff identify the music a resident with dementia may have preferred when s/he was young by asking family members and testing individual songs with the resident. Details of the second parallel trial conducted under this funding mechanism are registered under "R33AG057451_part2."**

The aims of this study are: 1. To use a train-the-trainer model to implement the intervention with ongoing monitoring of the program's adoption and acceptance by nursing home residents with dementia; 2. To estimate the impact of Music and Memory on agitated and aggressive behaviors; and 3. To examine factors associated with variation in providers' adherence to the implementation of Music and Memory.

ELIGIBILITY:
Inclusion Criteria for Nursing Homes:

* Owned by partnering health care corporations
* Medicare / Medicaid-certified
* Have at least 20 eligible residents

Inclusion Criteria for Residents in Eligible Nursing Homes

* Reside in eligible nursing home for last 90 days
* Have advanced dementia, defined by the presence of a dementia diagnosis and moderately or severely impaired daily decision-making

Exclusion Criteria for Nursing Homes:

* recent situations that may affect implementation (for example, bad state or federal quality assurance surveys, leadership turnover, or other competing demands)
* previous use of Music and Memory

Exclusion Criteria for Residents in Eligible Nursing Homes:

* dislikes music
* completely deaf

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1073 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mor, PhD, Principal Investigator — Brown University, School of Public Health
Locations (4):
- United States (4):
  - PruittHealth, Norcross, Georgia
  - Vetter Senior Living, Elkhorn, Nebraska
  - CommuniCare Terrapins Division, Blue Ash, Ohio
  - Good Samaritan Society, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conard RA, Baier RR, Sisti A, Dionne L, McCreedy EM. Resident and Nursing Home Factors Associated With Adherence to a Personalized Music Intervention: Secondary Analyses From Music & MEmory: A Pragmatic TRial for Nursing Home Residents With ALzheimer's Disease (METRIcAL). J Aging Res. 2025 May 2;2025:2679462. doi: 10.1155/jare/2679462. eCollection 2025. PMID 40352475
- [Derived] Davoodi NM, Dionne L, Mor V, McCreedy EM. Personalization of Reminiscence Therapies in the Nursing Home Setting: Lessons from an Embedded Pragmatic Trial of a Music Intervention. J Am Med Dir Assoc. 2023 Sep;24(9):1277-1278.e2. doi: 10.1016/j.jamda.2023.04.027. Epub 2023 Jun 2. No abstract available. PMID 37277100
- [Derived] McCreedy EM, Sisti A, Gutman R, Dionne L, Rudolph JL, Baier R, Thomas KS, Olson MB, Zediker EE, Uth R, Shield RR, Mor V. Pragmatic Trial of Personalized Music for Agitation and Antipsychotic Use in Nursing Home Residents With Dementia. J Am Med Dir Assoc. 2022 Jul;23(7):1171-1177. doi: 10.1016/j.jamda.2021.12.030. Epub 2022 Jan 14. PMID 35038407
- [Derived] Olson MB, McCreedy EM, Baier RR, Shield RR, Zediker EE, Uth R, Thomas KS, Mor V, Gutman R, Rudolph JL. Measuring implementation fidelity in a cluster-randomized pragmatic trial: development and use of a quantitative multi-component approach. Trials. 2022 Jan 15;23(1):43. doi: 10.1186/s13063-022-06002-8. PMID 35033176
- [Derived] McCreedy EM, Gutman R, Baier R, Rudolph JL, Thomas KS, Dvorchak F, Uth R, Ogarek J, Mor V. Measuring the effects of a personalized music intervention on agitated behaviors among nursing home residents with dementia: design features for cluster-randomized adaptive trial. Trials. 2021 Oct 7;22(1):681. doi: 10.1186/s13063-021-05620-y. PMID 34620193

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nursing home
Period: Overall Study
Arm/Group | Music and Memory | Usual Care
Started | 532; 27 nursing home | 541; 27 nursing home
Completed | 483; 27 nursing home | 493; 27 nursing home
Not Completed | 49; 0 nursing home | 48; 0 nursing home
Not completed — Death | 37 | 31
Not completed — Discharged | 10 | 14
Not completed — Not present in facility at followup | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music and Memory | Usual Care | Total
Number analyzed (Participants) | 483 | 493 | 976
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.8 (12.2) | 80.8 (12.3) | 80.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 327 | 349 | 676
  Male | 156 | 144 | 300
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 124 | 120 | 244
  White | 345 | 362 | 707
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 483 | 493 | 976
Cognitive function [Count of Participants; unit: Participants]
  Cognitively intact | 52 | 61 | 113
  Mildly impaired | 102 | 104 | 206
  Moderately impaired | 252 | 257 | 509
  Severely impaired | 77 | 71 | 148

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Agitated and Aggressive Behaviors (Staff Report)
Description: The tool used to interview staff about resident behaviors is the Cohen-Mansfield Agitation Inventory. Research staff interview a nursing staff member who knows the resident well to ask how frequently 29 agitated and/or aggressive behaviors occurred in the past week. There are seven response choices for each item, anchored from never (1) to several times per hour (7). Total scores on the Cohen-Mansfield Agitation Inventory range from 29 to 203, with higher scores representing more frequent agitated and/or aggressive behaviors. Adjusted mean overall scores will be compared for treatment and control populations.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
score on scale | 50.31 (1.35) | 48.04 (1.35)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = 1.33, 95% CI 2-sided [-1.37 to 4.03], Standard Error of Mean 1.38; Fixed effects: age, sex, race, activities of daily living score, cognitive function score, psychotic disorder, bipolar disease, depression, anxiety, dementia, antidepressant use, antianxietal use, antipsychotic use, corporation, time from Minimum Data Set (MDS) collection to Cohen-Mansfield Agitation Inventory (CMAI) score (exclusive to CMAI model), baseline Agitation and Reactive Behavior Scale (ARBS) (exclusive to CMAI model), baseline CMAI (exclusive to ARBS and ARBS-CMAI model), indicator of baseline/follow-up score, treatment group, interaction of baseline/follow-up measure, and treatment group. Random effects: random intercept for nursing home, random intercept for the interaction of baseline/follow-up measure and nursing home, random intercept for data collector (exclusive to CMAI model), and random intercept for individual

2. Secondary Outcome: Frequency of Verbal Agitated and Aggressive Behaviors (Direct Observation)
Description: The tool used to directly observe resident behaviors is the Agitation Behavior Mapping Instrument. Research staff observe residents for short intervals (3 minutes per observation) and record the number of times 14 specific verbally and physically agitated behaviors occurred (up to 10 times per observation). Ordinal outcomes quantify the number of physical and verbal agitated behaviors that occurred during the ABMI observations. The levels of these outcomes are None (0), Some (1 - 3) and Many (4 or more) observed behaviors.
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with behavior
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with behavior
  None | 0.80 [0.74 to 0.85] | 0.80 [0.74 to 0.85]
  Some | 0.13 [0.09 to 0.17] | 0.13 [0.10 to 0.17]
  Many | 0.08 [0.06 to 0.10] | 0.07 [0.03 to 0.09]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = 0.06, 95% CI 2-sided [0.03 to 0.09] — Reported estimation details pertain to the None category; The intention-to-treat (ITT) analysis used Bayesian multi-level multinomial logit models. All models adjust for resident baseline covariates, an individual-level effect to account for multiple observations for the same resident, and a facility level effect to account for variability in the outcomes for individuals residing in the same nursing homes. The reference category for the multinomial model for each outcome is "None". To address baseline differences in the proportion of individuals at each level of the ordinal outcomes between treatment and control groups, we report the marginal time by intervention interaction

3. Secondary Outcome: Frequency of Agitated and Aggressive Behaviors (Administrative Data)
Description: The Aggressive Behavior Scale is a 4-item measure describing the frequency of physical behavioral symptoms directed toward others; verbal behavioral symptoms directed toward others; other behavioral symptoms not directed toward others; and behaviors related to resisting necessary care. For each item, frequency in the past week is reported as: behavior not exhibited (0); behavior occurred 1-3 days (1); behavior occurred 4-6 days (2); or behavior occurred daily (3). The Aggressive Behavior Scale ranges from 0 to 12, with higher scores indicating more frequent agitated and/or aggressive behaviors. Mean total scores will be compared for treatment and control populations.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
score on a scale | 0.42 (0.08) | 0.40 (0.08)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; Marginal Interaction Effect = -0.11, 95% CI 2-sided [-0.30 to 0.08], Standard Error of Mean 0.10; Fixed effect covariates: age, sex, race, activities of daily living score, cognitive function score, psychotic disorder, bipolar disease, depression, anxiety, dementia, antidepressant use, antianxietal use, antipsychotic use, nursing home corporation, time from Minimum Data Set (MDS) collection to Cohen-Mansfield Agitation Inventory (CMAI) score (exclusive to CMAI model), baseline Agitation and Reactive Behavior Score (ARBS) (exclusive to CMAI model), baseline CMAI (exclusive to ARBS and ARBS-CMAI model), indicator of baseline/follow-up score, treatment group, interaction of baseline/follow-up measure, and treatment group. Random effects: random intercept for nursing home, random intercept for the interaction of baseline/follow-up measure and nursing home, random intercept for data collector (exclusive to CMAI model), and random intercept for individual

4. Secondary Outcome: Antipsychotic Use
Description: Any antipsychotic use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
adjusted percentage of participants | 26.2 (1.4) | 29.6 (1.3)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -3.61, 95% CI 2-sided [-7.22 to 0.00], Standard Error of Mean 1.85; Variables included in the model: baseline medication use, age, sex, race, activities of daily living score, cognitive function score, psychotic diagnosis, depression, anxiety, dementia, asthma, agitation and reactive behavior (ARBS) score, date of assessment, treatment group, and facility-level random effect

5. Secondary Outcome: Antianxietal Use
Description: Any antianxietal use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
adjusted percentage of participants | 20.8 (1.5) | 24.3 (1.7)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -3.47, 95% CI 2-sided [-7.55 to 0.06], Standard Error of Mean 2.08; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Antidepressant Use
Description: Any antidepressant use in the past week and days of use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Measure type of mean is chosen based on adjusted percentage with standard errors from a multilevel, difference in difference regression models.
Time Frame: 4-months
Measure: Mean (Standard Error); unit: adjusted percentage of participants
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
adjusted percentage of participants | 57.5 (1.5) | 58.8 (1.5)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -1.26, 95% CI 2-sided [-5.28 to 2.76], Standard Error of Mean 2.05; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Hypnotic Use
Description: Any hypnotic use in the past week, based on Minimum Data Set (standardized assessment of nursing home residents). Comparison of percent with any use will be compared for treatment and control populations.
Time Frame: 4-months
Measure: Number; unit: unadjusted percentage of participants
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
unadjusted percentage of participants | 0.83 | 1.22

8. Secondary Outcome: Depression
Description: The Patient Health Questionnaire is a 9-item screening assessment for depression severity. For each item, respondents indicate the frequency of the symptom in the past 2 weeks using the following choices: never or one day (0); 2-6 days (1); 7-11 days (2); or 12-14 days (3). Total scores range from 0 to 27, with higher scores indicating more frequent depressive symptoms. Average total scores will be compared for treatment and control populations.
Time Frame: 4-months
Population: Participants dropped from analysis if missing PHQ-9 score at baseline or followup
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 469 | 479
score on a scale | 2.09 (0.33) | 2.30 (0.33)
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -0.22, 95% CI 2-sided [-1.14 to 0.70]; Multilevel regression with covariates' adjustments was used to estimate the impact of the resident being in a treatment versus control nursing home on depressive symptoms

9. Secondary Outcome: Frequency of Physical Agitated and Aggressive Behaviors (Direct Observation)
Description: The tool used to directly observe resident behaviors is the Agitation Behavior Mapping Instrument. Research staff observe residents for short intervals (3 minutes per observation) and record the number of times 14 specific verbally and physically agitated behaviors occurred (up to 10 times per observation). We report the proportion of participants with no behaviors, some behaviors (1-3 ), many behaviors (4+)
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with behavior
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with behavior
  None | 0.85 [0.80 to 0.90] | 0.90 [0.85 to 0.94]
  Some | 0.12 [0.08 to 0.17] | 0.09 [0.06 to 0.13]
  Many | 0.03 [0.02 to 0.04] | 0.01 [0.01 to 0.02]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = 0.00, 95% CI 2-sided [-0.03 to 0.02] — Reported estimation details pertain to the None category; The intention-to-treat (ITT) analysis used Bayesian multi-level multinomial logit models to analyze the effect that being in a treatment versus control nursing home had on the behaviors of nursing home residents. All models adjust for resident baseline covariates and the activity status of a resident during an observation. In addition, they include an individual-level effect to account for multiple observations for the same resident, and a facility level effect to account for variability in the outcomes for individuals residing in the same nursing homes. To address baseline differences in the proportion of individuals at each level of the ordinal outcomes between treatment and control groups, we report the marginal time by intervention interaction

10. Secondary Outcome: Observed Pleasure
Description: The Observed Emotion Rating Scale is completed by a trained observer to document duration of five observed emotional states (pleasure, anger, anxiety / fear, sadness, and general alertness) during short observations (3 minutes per observation). For each emotional state, the researcher indicates whether or not the emotion was observed: never (1); less than 16 seconds (2); 16-59 seconds (3); 1-2 minutes (4); or 3+ minutes (5). Total scores range from 5 to 25, with higher scores indicating greater duration of observed emotion. We report the proportion of participants with any observed emotion during the structured observations after four months of follow-up.
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with behavior
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with behavior | 0.36 [0.30 to 0.43] | 0.29 [0.24 to 0.35]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = 0.05, 95% CI 2-sided [0.02 to 0.07]; The intention-to-treat (ITT) analysis used Bayesian multi-level multinomial logit models to analyze the effect that being in a treatment versus control nursing home had on the moods of nursing home residents. All models adjust for resident baseline covariates and the activity status of a resident during an observation. In addition, they include an individual-level effect to account for multiple observations for the same resident, and a facility level effect to account for variability in the outcomes for individuals residing in the same nursing homes. We report the marginal time by intervention interaction

11. Secondary Outcome: Observed Anger
Description: The Observed Emotion Rating Scale is completed by a trained observer to document duration of five observed emotional states (pleasure, anger, anxiety / fear, sadness, and general alertness) during short observations (3 minutes per observation). For each emotional state, the researcher indicates whether or not the emotion was observed: never (1); less than 16 seconds (2); 16-59 seconds (3); 1-2 minutes (4); or 3+ minutes (5). Total scores range from 5 to 25, with higher scores indicating greater duration of observed emotion. Average observed emotion scores will be compared for treatment and control populations. We report the proportion of participants with any observed anger during observations after four months of followup.
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with emotion
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with emotion | 0.04 [0.03 to 0.06] | 0.03 [0.02 to 0.04]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = -0.01, 95% CI 2-sided [-0.03 to 0.01]; [other analysis details as in outcome 10, analysis 1]

12. Secondary Outcome: Observed Sadness
Description: The Observed Emotion Rating Scale is completed by a trained observer to document duration of five observed emotional states (pleasure, anger, anxiety / fear, sadness, and general alertness) during short observations (3 minutes per observation). For each emotional state, the researcher indicates whether or not the emotion was observed: never (1); less than 16 seconds (2); 16-59 seconds (3); 1-2 minutes (4); or 3+ minutes (5). Total scores range from 5 to 25, with higher scores indicating greater duration of observed emotion. Average observed emotion scores will be compared for treatment and control populations. We report the proportion of participants any sadness observed during structured observations after four months of follow-up
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with emotion
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with emotion | 0.07 [0.05 to 0.11] | 0.06 [0.04 to 0.10]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; average marginal effect = -0.01, 95% CI 2-sided [-0.04 to 0.01]; [other analysis details as in outcome 10, analysis 1]

13. Secondary Outcome: Observed Alertness
Description: The Observed Emotion Rating Scale is completed by a trained observer to document duration of five observed emotional states (pleasure, anger, anxiety / fear, sadness, and general alertness) during short observations (3 minutes per observation). For each emotional state, the researcher indicates whether or not the emotion was observed: never (1); less than 16 seconds (2); 16-59 seconds (3); 1-2 minutes (4); or 3+ minutes (5). Total scores range from 5 to 25, with higher scores indicating greater duration of observed emotion. Average observed emotion scores will be compared for treatment and control populations. We report the proportion of participants with any observed alertness during structured observations after four months of followup
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with emotion
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with emotion | 0.78 [0.74 to 0.82] | 0.76 [0.72 to 0.80]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = 0.01, 95% CI 2-sided [-0.02 to 0.03]; [other analysis details as in outcome 10, analysis 1]

14. Secondary Outcome: Observed Anxiety
Description: The Observed Emotion Rating Scale is completed by a trained observer to document duration of five observed emotional states (pleasure, anger, anxiety / fear, sadness, and general alertness) during short observations (3 minutes per observation). For each emotional state, the researcher indicates whether or not the emotion was observed: never (1); less than 16 seconds (2); 16-59 seconds (3); 1-2 minutes (4); or 3+ minutes (5). Total scores range from 5 to 25, with higher scores indicating greater duration of observed emotion. Average observed emotion scores will be compared for treatment and control populations. We report the proportion of participants with any observed anxiety during structured observations after four months of follow-up
Time Frame: 4-months
Measure: Number (95% Confidence Interval); unit: proportion of participants with emotion
Arm/Group | Music and Memory | Usual Care
Number analyzed (Participants) | 483 | 493
proportion of participants with emotion | 0.12 [0.08 to 0.17] | 0.13 [0.08 to 0.18]
Statistical Analysis 1: Comparison: Music and Memory vs Usual Care; Test type: Superiority; p < 0.05, Differences-in-Differences regression; marginal interaction effect = -0.02, 95% CI 2-sided [-0.05 to 0.01]; The intention-to-treat (ITT) analysis used Bayesian multi-level multinomial logit models to analyze the effect that being in a treatment vs. control NH had on the behaviors and moods of NH residents. The models were implemented separately for each mood. All models adjust for resident baseline covariates and the activity status of a resident during an observation. In addition, they include an individual-level effect to account for multiple observations for the same resident, and a facility level effect to account for variability in the outcomes for individuals residing in the same nursing homes. To address baseline differences in the proportion of individuals at each level of the ordinal outcomes between treatment and control groups, we report the marginal time by intervention interaction. We will refer to this estimand as the marginal interaction effect (MIE), which is sometimes known as the Difference in Differences estimand

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Music and Memory | Usual Care
All-Cause Mortality (participants affected / at risk) | 37/532 | 31/541
Serious Adverse Events (participants affected / at risk) | 0/532 | 0/541
Other Adverse Events (participants affected / at risk) | 0/532 | 0/541

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03821844/Prot_SAP_000.pdf